CLINICAL TRIAL: NCT04955860
Title: Evaluation of First Molar Inclinations and Dental Arch Parameters in Individuals With Bilateral Posterior Crossbite at Different Age Periods
Brief Title: Evaluation of First Molar Inclinations and Transverse Arch Width in Individuals With Posterior Crossbite
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Taner OZTURK, DDS, MS, Lecturer, TC Erciyes University
Other Study IDs: 2020/44
Record Dates: First submitted 2021-07-05; First posted 2021-07-09 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Crossbite (Anterior) (Posterior); Dental Malocclusion; Maxillary Anomaly
Keywords: posterior crossbite; dental model analysis; molar inclination; dental arch parameter
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Data of cast plaster model scans of the lower and upper jaws obtained from individuals for routine treatment procedures were obtained and stored digitally.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: Individuals with bilateral posterior crossbite will be included.
  Interventions: Other: Dental model analysis
- Control Group: Individuals with no anterior and/or posterior crossbite and transversal malocclusion will be included.
  Interventions: Other: Dental model analysis

INTERVENTIONS:
Other: Dental model analysis — No interventional treatment intervention will be made for individuals. Digital dental models taken for orthodontic recording will be examined.

SUMMARY:
This study aims to evaluate and compare the inclination of the lower and upper permanent first molars and the transversal width of the lower and upper jaws in individuals of different age groups to evaluate whether the existing anomaly at different ages in individuals with a bilateral posterior crossbite. For this reason, first molar tooth inclination and lower and upper jaw transversal width will be evaluated in adolescent and post-adolescent individuals with a bilateral posterior crossbite.

DETAILED DESCRIPTION:
The maxillary dental arch covers the mandibular arch in every space like a box cover in normal occlusion. The transversal disappearance of this relationship is called a crossbite. If this deformity occurs between posterior group teeth, it is defined as a posterior crossbite. In other words, in posterior crossbite, while the teeth are in centric occlusion, the vestibule tubercles of the upper posterior teeth come into contact with the central fossa of the lower posterior teeth. This occlusal discrepancy may concern only one tooth, or it may involve multiple teeth or all teeth. A posterior crossbite can be observed unilaterally or bilaterally and is usually caused by insufficient width of the upper jaw compared to the lower jaw.

Crossbite; stated that it is a term used for the abnormal buccal, labial, or lingual relations of the lower and upper jaw teeth or tooth groups when the lower and upper dental arches are in the closing state. Crossbite is divided into two groups as anterior and posterior crossbite according to the region in the mouth. Anterior crossbite indicates malocclusion of the jaws and/or dental arches in the sagittal direction, while posterior crossbite indicates malocclusion in the transversal direction. Posterior crossbite is defined as the contact of the buccal tubercles of the posterior maxillary teeth with the lingual tubercles of the opposite mandibular teeth. This anomaly can be seen unilaterally or bilaterally and may involve one or more teeth. In addition, although the canines were anterior teeth before, these teeth were included in the posterior region while expressing posterior crossbite. A posterior crossbite can be seen in the primary, mixed, and permanent dentition period.

Posteroanterior (PA) cephalograms are the most readily available and reliable diagnostic tool for the radiological identification and evaluation of transversal irregularities. Traditionally, orthodontists have focused on two-dimensional lateral cephalograms; however, treatment is done in all three planes. A planar assessment of the transverse space cannot be made unless the PA cephalogram is analyzed. Typically, standard PA cephalograms were not used as part of routine diagnostic recordings. However, PA radiographs should be added as an additional recording material in individuals with a posterior crossbite.

Digital radiographs and digital photographs are becoming the norm in orthodontic records. Recent developments also include electronic working models. Because the medical and dental anamnesis, digital photos, radiographs, and all treatment notes were in digital format have become desirable to obtain digital study models. Dental cast models have a long and proven history in orthodontics. It has become the "gold standard" in orthodontics with many advantages, from cast models that can be mounted on an articulator for a three-dimensional study, from routine dental examination to ease of manufacture, cheapness, and ease of measurement. Digital operating models offer advantages that include storage and reassessment, ease of cross-transmission, and possibly equal or better diagnostic capabilities. In addition, linear dental anatomical measurements were obtained from plaster and digital models, while Bolton analysis was performed on the cast and digital models.

At the beginning of the treatment, dental plaster models obtained from the lower and upper jaw dimensions will be scanned with a three-dimensional model scanning device (3 Shape R700 3D Scanner, 3 Shape A/S, Copenhagen, Denmark). Scanned models will be analyzed with the 3Shape Orthoanalyzer program (3Shape A/S, Copenhagen, Denmark). A point will be placed on the distal, facial, mesial, and lingual surfaces of each tooth, from the right first permanent molar to the left first permanent molar in the same arch. These points will be chosen by the rules established by Moyers et al. and Brust and McNamara to determine the geometric center of each tooth, the tooth center. This point provides a broader arc width measurement because it will eliminate the effect of tooth rotation. After cast rotation, the first molars' facial and lingual cusp crests will be selected to assess molar tooth tilt and angulation. An inclination below 180 degrees indicates that the molars are inclined buccally, while values above 180 degrees indicate that these teeth are inclined lingually.

Dental arch width measurements will be measured between the following teeth: permanent canines, first premolars, second premolars, and permanent first molars. Arch width will be evaluated with two sets of measurements: the distance from the lingual point of the selected tooth to the similar point on its antimere and between the centroid and antimer of a tooth.

The arch depth shall be measured as the distance from the midpoint between the facial surfaces of the central incisors to the tangent line to the mesial surfaces of the first permanent molars. Arch circumference will be determined by summing the segments between the points of contact from the mesial surface of the first permanent molar to the mesial surface of the opposite first permanent molar.

ELIGIBILITY:
Inclusion Criteria:

* For the Working Group;

  1. Absence of a syndrome or disease affecting the craniofacial and general systemic condition
  2. Patients who have applied for treatment due to the need for orthodontic treatment
  3. Adequate radiographic and three-dimensional dental model records before treatment
  4. Bilateral posterior crossbite
  5. Absence of anterior crossbite
  6. Absence of loss of lower and upper first permanent molars and eruption of all 4 permanent molars
* For the Control Group;

  1. Absence of a syndrome or disease affecting the craniofacial and general systemic condition
  2. Patients who have applied for treatment due to the need for orthodontic treatment
  3. Adequate radiographic and three-dimensional dental model records before treatment
  4. Absence of posterior and anterior crossbite
  5. Absence of loss of lower and upper first permanent molars and eruption of all 4 permanent molars

Exclusion Criteria:

1. Presence of a syndrome and disease affecting the craniofacial and general systemic condition
2. Absence of radiographic and dental model records
3. Losing any of the lower or upper permanent first molars
4. Presence of anterior crossbite

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Differences between male and female individuals will also be evaluated separately for each group and parameter.
Study Population: Individuals with and without posterior crossbite who applied for orthodontic treatment
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Mandibular and maxillary first molar positions | At the beginning of the examination, it will be evaluated as an average of 10 minutes for each patient's lower and upper jaw.
  The inclinations of the lower and upper permanent first molars in the frontal plane will be evaluated.
Dimensions of the upper dental arch in the transverse direction | At the beginning of the examination, it will be evaluated as an average of 15 minutes for each patient's maxilla.
  The distances of the right and left permanent canines, first and second premolars, and permanent first molars transversely to each other in the upper jaw of each patient will be evaluated. In addition, dental arch perimeter and dental arch depth will be evaluated.
Dimensions of the lower dental arch in the transverse direction | At the beginning of the examination, it will be evaluated as an average of 15 minutes for each patient's mandible.
  The distances of the right and left permanent canines, first and second premolars, and permanent first molars transversely to each other in the upper jaw of each patient will be evaluated. In addition, dental arch perimeter and dental arch depth will be evaluated.
Evaluation of the transverse dimensions of the lower and upper jaws between different age groups | At the beginning of the examination, it will be evaluated as an average of 25 minutes for each patient's mandible.
  The differences between the periods of different age groups (12-14 years, 14-16 years and 16-18 years) will also be evaluated separately for each group and parameter.

SECONDARY OUTCOMES:
Evaluation of the transverse dimensions of the lower and upper jaws between the sexes | At the beginning of the examination, it will be evaluated as an average of 25 minutes for each patient's mandible.
  Differences between male and female individuals will also be evaluated separately for each group and parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Yagci, DDS, PhD, Study Director — Erciyes University, Faculty of Dentistry, Department of Orthodontics; Sabri I Ramoglu, DDS, PhD, Study Chair — Altinbas University, Faculty of Dentistry, Department of Orthodontics
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical restrictions.

REFERENCES:
- [Background] McNamara JA Jr, Baccetti T, Franchi L, Herberger TA. Rapid maxillary expansion followed by fixed appliances: a long-term evaluation of changes in arch dimensions. Angle Orthod. 2003 Aug;73(4):344-53. doi: 10.1043/0003-3219(2003)0732.0.CO;2. PMID 12940553
- [Background] da Silva Filho OG, Ferrari Junior FM, Okada Ozawa T. Dental arch dimensions in Class II division 1 malocclusions with mandibular deficiency. Angle Orthod. 2008 May;78(3):466-74. doi: 10.2319/022307-89.1. PMID 18416613
- [Background] McNamara JA Jr. Early intervention in the transverse dimension: is it worth the effort? Am J Orthod Dentofacial Orthop. 2002 Jun;121(6):572-4. doi: 10.1067/mod.2002.124167. No abstract available. PMID 12080303